CLINICAL TRIAL: NCT03677336
Title: Oral Dydrogesterone Versus Micronized Vaginal Progesterone for Luteal Phase Support in In Vitro Fertilisation (IVF)/ IntraCytoplasmic Sperm Injection (ICSI): Pharmacokinetics and the Impact on the Endometrium, the Microbiota of the Genital Tract and the Peripheral Immunology. Double Blind Crossover Study.
Brief Title: Oral Dydrogesterone (OD) Versus Micronized Vaginal Progesterone (MVP) for Luteal Phase Support (LPS) in IVF/ICSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CRG UZ Brussel (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Abbott (Industry); KU Leuven (Other)
Responsible Party: Principal Investigator, Mackens Shari, Principal investigator, CRG UZ Brussel
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DYDRA001; 2018-000105-23 (EudraCT Number)
Record Dates: First submitted 2018-09-04; First posted 2018-09-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Infertility, Female; Infertility; Genital Diseases, Male; Genital Diseases, Female; Progesterone; Dydrogesterone; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Physiological Effects of Drugs; Progestins
MeSH Terms: conditions — Infertility, Female; Infertility; Genital Diseases, Male; Genital Diseases, Female | interventions — Dydrogesterone; Progesterone; Utrogestan

STUDY DESIGN:
Intervention Model Description: A randomised, cross-over, double blind double dummy study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded and packaged medication will be provided to the investigational site and dispensed to the participants. The participants, their treating physicians and the investigators will be blinded for the randomization of subjects to the treatment groups. Of both treatment medications, OD and MVP, a placebo version will be available and administered in both oocyte donation cycles. The medication will be given in a double blind double dummy fashion. All the tablets and capsules will be identical in appearance, shape, smell and taste, and packaged in the proper proportion to assure desired dosages and maintenance of the blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group l: 1st cycle MVP/placebo OD (Other): 2 cycles of controlled ovarian stimulation, dual triggering, oocyte retrieval (OR) and LPS, with an interval period of 2 to 12 months. The only difference of the second cycle being the other LPS study medication as compared to the first cycle.
  * 1st cycle: Start on day of oocyte retrieval (OR) (=d1): Dydrogesterone Oral Tablet 10 mg 3 times daily + Placebo micronized vaginal progesterone 200 mg capsules 3 times daily, for 8 days.
  * 2nd cycle: Start on day of oocyte retrieval (OR) (=day 1): 'Micronized Progesterone 200 mg intravaginal capsules 3 times daily + placebo 'Dydrogesterone Oral Tablet 10 mg 3 times daily, for 8 days.
  Interventions: Drug: Dydrogesterone Oral Tablet; Drug: Micronized progesterone; Drug: Placebo Dydrogesterone oral tablet; Drug: Placebo Micronized progesterone
- Group ll: 1st cycle placebo MVP/OD (Other): 2 cycles of controlled ovarian stimulation, dual triggering, oocyte retrieval (OR) and LPS, with an interval period of 2 to 12 months. The only difference of the second cycle being the other LPS study medication as compared to the first cycle.
  * 1st cycle: Start on day of oocyte retrieval (OR) (=day 1): Micronized Progesterone 200 mg intravaginal capsules 3 times daily + placebo Dydrogesterone Oral Tablet 10 mg 3 times daily, for 8 days.
  * 2nd cycle: Start on day of oocyte retrieval (OR) (=day 1): Dydrogesterone Oral Tablet 10 mg 3 times daily + Placebo micronized progesterone 200 mg intravaginal capsules 3 times daily, for 8 days.
  Interventions: Drug: Dydrogesterone Oral Tablet; Drug: Micronized progesterone; Drug: Placebo Dydrogesterone oral tablet; Drug: Placebo Micronized progesterone

INTERVENTIONS:
Drug: Dydrogesterone Oral Tablet — Tablet, oral, 10 mg, 3 times daily, starting on the day of oocyte retrieval in the morning and during 8 days
  Other Names: OD; Duphaston
Drug: Micronized progesterone — Capsule, vaginal, 200 mg, 3 times daily, starting on the day of oocyte retrieval in the morning and during 8 days
  Other Names: MVP; Utrogestan
Drug: Placebo Dydrogesterone oral tablet — Tablet, indistinguishable from dydrogesterone oral tablet
  Other Names: Placebo OD
Drug: Placebo Micronized progesterone — Capsule, indistinguishable from micronized vaginal progesterone capsules
  Other Names: Placebo MVP

SUMMARY:
Female inability to conceive a child. The purpose of this prospective randomized, double-blinded, double dummy, two-arm cross-over study is to investigate the difference on histological, transcriptional and immunological level in endometrium between 3x10mg Dydrogesterone oral tablets and 3x200 mg Micronized progesterone intravaginal capsules for the luteal support in egg cell donors. Beside that, the pharmacokinetics, the impact on the peripheral immunology (by blood sampling) and the microbiota (by genital swabs) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donor candidates
* Regularly cycling
* BMI ≥18 and ≤ 29 kg/m2
* Signed informed consent
* Non-smokers.
* AMH <7,53 and >1,18 ng/mL (90th and 10th percentile for healthy women aged 25-29 according to the used Elecsys® AMH kit by Roche)
* PRL, T and TSH within the normal limits for the clinical laboratory, or considered not clinically significant by the investigator within 6 months prior or at screening

Exclusion Criteria:

* Intra-uterine device
* Previous enrollment
* Evidence of cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatologic/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurologic/psychiatric, allergy, recent major surgery (< 3 months), or other relevant diseases as revealed by history, physical examination and/or laboratory assessments which could limit participation in or completion of the study
* Acute urogenital disease during the course of the study
* Known allergic reactions to progesterone / dydrogesterone products (active substance or to any of the excipients)
* Intake of any experimental drug or any participation in any other clinical trial within 30 days prior to study start.
* Mental disability or any other lack of fitness, in the investigator's opinion, to preclude subjects in or to complete the study.
* Current or recent substance abuse, including alcohol and tobacco (patients who stopped tobacco usage at least 3 months prior to screening visit would be allowed)
* Refusal or inability to comply with the requirements of the study protocol for any reason, including scheduled clinic visits and laboratory tests.
* Known or suspected progestogen dependent neoplasms (e.g. meningioma)
* Serum progesterone level >1.5 ng/mL at ovulation triggering

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Molecular endometrial level using illumina RNA-seq | On the eight day (at 8am) of LPS intake
  To study the difference of OD versus MVP as LPS after controlled ovarian stimulation (COS) on the molecular endometrial level using Illumina RNA-seq on endometrial derived single cell suspensions
Molecular endometrial level using immunohistochemistry | On the eight day (at 8am) of LPS intake
  To study the difference of OD versus MVP as LPS after controlled ovarian stimulation (COS) on the molecular endometrial level using immunohistochemistry on endometrial derived single cell suspensions
Molecular endometrial level using flow cytometry | On the eight day (at 8am) of LPS intake
  To study the difference of OD versus MVP as LPS after controlled ovarian stimulation (COS) on the molecular endometrial level using flow cytometry on endometrial derived single cell suspensions

SECONDARY OUTCOMES:
Difference in pharmacokinetic profile: Progesterone: AUC0-τ | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: AUC0-t | On the first day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: Cmax | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: tmax | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: Ctrough | On the eight day of LPS intake: 1 hour before morning dose.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: λz | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: t1/2 | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: CL/F | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Progesterone: Vz/F | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: AUC0-τ | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: ratios of AUC0-τ of dydrogesterone and DHD | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: AUC0-t | On the first day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: ratios of AUC0-t of dydrogesterone and DHD | On the first day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: Cmax | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: ratios of Cmax of dydrogesterone and DHD | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: tmax | On the first and eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: Ctrough | On the eight day of LPS intake: 1 hour before morning dose.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: λz | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: t1/2 | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: CL/F | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in pharmacokinetic profile: Dydrogesterone and 20α-dihydrodydrogesterone: Vz/F | On the eight day of LPS intake: 1 hour before morning dose, 0.5 hour, 1 hour, 1 hour 30, 2 hours, 2 hours 30, 3 hours, 4 hours, 5 hours post-dose. One blood sample on the 9th, 10th and 11th day.
  using Liquid Chromatography with tandem Mass Spectrometry (LC-MS/MS)
Difference in peripheral immunology | On the first and eight day of LPS intake, 1hour before morning dose at 9 am.
  To study the effects of OD versus MVP on the peripheral immunology (using flow cytometry to investigate T regulatory and T effector cells derived from peripheral blood)
Difference in microbiota in the female genital tract | On the first and eight day of LPS intake, 1 hour before morning dose at 9 am.
  by cervical swab, a vaginal swab (posterior fornix) and an intra-uterine sample using an empty embryo catheter. Evaluation using 16S rRNA amplicon sequencing - Illumina miSeq

CONTACTS AND LOCATIONS:
Overall Officials: Herman Tournaye, PhD, MD, Principal Investigator — Head of department CRG
Locations (1):
- Centrum voor Reproductieve Geneeskunde, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tournaye H, Sukhikh GT, Kahler E, Griesinger G. A Phase III randomized controlled trial comparing the efficacy, safety and tolerability of oral dydrogesterone versus micronized vaginal progesterone for luteal support in in vitro fertilization. Hum Reprod. 2017 May 1;32(5):1019-1027. doi: 10.1093/humrep/dex023. PMID 28333318